CLINICAL TRIAL: NCT00498108
Title: An Open-label Extension Trial to Investigate the Safety and Tolerability of Long-term Treatment With Transdermal Rotigotine in Subjects With Idiopathic Restless Legs Syndrome
Brief Title: Phase 3 Open-label Extension Trial With Rotigotine in Idiopathic Restless Legs Syndrome Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SP0791; EudraCT Number: 2005-002611-25
Record Dates: First submitted 2007-07-06; First posted 2007-07-09 (Estimated); Last update posted 2014-09-25 (Estimated); Status verified 2009-09

CONDITIONS: Idiopathic Restless Legs Syndrome
Keywords: Rotigotine; Restless Legs Syndrome
MeSH Terms: conditions — Restless Legs Syndrome | interventions — rotigotine

INTERVENTIONS:
Drug: Rotigotine

SUMMARY:
This is a multicenter, open-label trial to assess safety and tolerability of rotigotine in subjects with idiopathic Restless Legs Syndrome (RLS), administered at an optimal dose for up to 1 year in subjects who previously participated in SP790 (6-month pivotal trial) or SP794 (sleep lab trial). Subjects who successfully completed the Maintenance Period and the Taper Period of SP790 or SP794 are allowed to enroll in this trial.

ELIGIBILITY:
Inclusion Criteria:

* Subject completed the Maintenance Period and Taper Period of SP790 or SP794

Exclusion Criteria:

* Subject has an ongoing serious adverse event (SAE) from SP790 or SP794 that is assessed to be related to the trial medication by the investigator and/or the sponsor.
* Subject has any medical or psychiatric condition that, in the opinion of the investigator, can jeopardize or would compromise the subject's ability to participate in this trial

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 341 (Actual)
Dates: Start 2006-01; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Adverse events, changes in laboratory tests, vital signs, physical and neurological examination, menstrual and sexual function, 12-lead ECGs. Subject's rating of daytime sleepiness, global subject rating of tolerability

SECONDARY OUTCOMES:
Change in the International Restless Legs Scale (IRLS) sum score, in CGI Items 1 and 2-3, in RLS-6 Rating Scales. IRLS Responder | from Baseline at the end of the Maintenance Period

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — UCB Pharma
Locations (1):
- Kassel, Germany